CLINICAL TRIAL: NCT07002190
Title: The Effect of Education Given Before Port Catheter Infusion on Infusion Related Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Yekta Demirsoy, nurse, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-23
Record Dates: First submitted 2025-05-10; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Port-A-Cath
Keywords: Pain; Anxiety; Education; Nursing; Port catheter
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The Experimental group period with the support of visual education material
  Interventions: Other: Watching an animation video
- Control Group (No Intervention): The control group will take rutin patient çare.

INTERVENTIONS:
Other: Watching an animation video — education
  Arms: Experimental group

SUMMARY:
Pain, anxiety, anxiety and changes in vital signs are observed in patients during needle insertion into the port catheter.Patients and their relatives should be informed by nurses to eliminate these problems and to provide more comfortable infusion to patients.However, studies on the care process for the symptoms that occur before port catheter infusion are limited in the literature.The thesis study planned for this purpose will be carried out to determine the effect of the training given before port catheter infusion on infusion-related symptoms.The research will be conducted as pretest-posttest, randomised controlled.Oncology-Hematology Services and Chemotherapy Unit of Karadeniz Technical University Farabi Hospital.The sample of the study will be determined by simple randomisation method and 64 patient will be included in the study.The data of the study will be collected by Patient Descriptive Information Form, Visual Analogue Scale and State and Trait Anxiety Scale, Vital Signs Follow-up Chart.

ELIGIBILITY:
Inclusion Criteria:

* Having a port catheter
* The patient has no previous experience with a port catheter,
* The patient will receive an infusion from a port catheter for the first time,
* The patient's age range is between 18-70,
* The patient is literate,
* Volunteering to participate in the study,
* The patient will receive training from the training material for the first time.

Exclusion Criteria:

* Those with communication, hearing and vision problems,
* Those with any psychiatric disorder,
* Those who used any analgesic medication at least 8 hours before

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Identifying Information Form | 1 day
  This form, which was created by the researchers by reviewing the relevant literature, consists of 11 questions evaluating the descriptive characteristics of the patients the number of port catheter needle insertions and the information status about the port catheter.

SECONDARY OUTCOMES:
State and Trait Anxiety Scale | 2 day
  The scale, which is in the z-type evaluation type, consists of 2 subscales in the four-point Likert type and a total of 40 items. The answer options collected in four classes in the State Anxiety Scale include the expressions (1) Never, (2) A Little, (3) A Lot, (4) Completely, while the Trait Anxiety Scale includes four classes and includes the expressions (1) Almost never, (2) Sometimes, (3) A Lot, (4) Almost always.
Symptom chart | 2 day
  This form is used to measure patients' vital signs, pain during the procedure, and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şule Bıyık Bayram, Assoc. Prof. Dr., Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT07002190/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT07002190/ICF_001.pdf